CLINICAL TRIAL: NCT02559635
Title: Does Bowel Stimulation Before Loop Ileostomy Closure Reduce Postoperative Ileus? A Multicenter Randomized Controlled Trial
Brief Title: Does Bowel Stimulation Before Loop Ileostomy Closure Reduce Postoperative Ileus?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Collaborators: Montreal General Hospital (Other); North York General Hospital (Other); St. Mary's General Hospital (Unknown); Rush University Medical Center (Other); North Shore Hospital, Waitemata District Health Board (Unknown)
Responsible Party: Principal Investigator, Dr. Marylise Boutros, Assistant Professor, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JGH-06-2015
Record Dates: First submitted 2015-07-14; First posted 2015-09-24 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Ileus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No bowel stimulation (No Intervention): Patients undergoing loop ileostomy closures without having had bowel stimulation beforehand
- Bowel stimulation (Experimental): Patients undergoing loop ileostomy closures having undergone bowel stimulation beforehand
  Interventions: Procedure: Bowel stimulation; Drug: Nestle Resource

INTERVENTIONS:
Procedure: Bowel stimulation — Stimulation will be performed daily on an outpatient basis for the two weeks (ten business days) prior to ileostomy closure by a trained research assistant. The efferent limb of the ileostomy loop will be canalized with an 18 Fr Foley catheter and infused with a solution comprising of 500mL of normal saline mixed with 30g of a thickening-agent (Nestle Resource). It will be prepared in five 100mL syringes and administered slowly over 20 minutes.
  Arms: Bowel stimulation
Drug: Nestle Resource — Stimulation will be performed daily on an outpatient basis for the two weeks (ten business days) prior to ileostomy closure by a trained research assistant. The efferent limb of the ileostomy loop will be canalized with an 18 Fr Foley catheter and infused with a solution comprising of 500mL of normal saline mixed with 30g of a thickening-agent (Nestle Resource). It will be prepared in five 100mL syringes and administered slowly over 20 minutes.
  Arms: Bowel stimulation

SUMMARY:
Postoperative ileus is the most commonly observed morbidity following ileostomy closure. Studies have previously demonstrated that the defunctionalized bowel of a loop ileostomy undergoes a series of functional and structural changes. It has been hypothesized that these changes may contribute to the development of postoperative ileus, and that stimulating the distal limb of a loop ileostomy prior to closure may functionally prepare the excluded bowel for intestinal transit.

The purpose of the multicenter, randomized controlled trial is to determine the impact of preoperative stimulation of the distal limb of a loop ileostomy on postoperative ileus.

DETAILED DESCRIPTION:
Low anterior resection with total mesorectal excision is the standard operative treatment for mid and some low rectal cancers.The most dreaded and morbid complication of this procedure is anastomotic leak,with a varied incidence of 3-32%,and which can result in pelvic abscess and sepsis,re-operation,and death.The creation of a loop ileostomy is the only measure proven to reduce the morbidity and septic complications of anastomotic leakage. With the current trend towards sphincter-preserving surgery and the performance of ultra-low anastomoses for low rectal cancers, anastomotic dehiscence is increasingly being observed.That, in addition to the frequent use of neoadjuvant radiotherapy has contributed to a greater use of diverting ostomies. Furthermore, the use of a protective loop ileostomy is not limited to oncologic surgeries, and is often performed during colonic resection for complicated diverticular disease.

However, the formation of a loop ileostomy comes at a price as it requires a second surgery typically 12 weeks after the initial operation to restore intestinal continuity. The incidence of complications following ileostomy closure is certainly not negligible, at a highly variable range of 11-45%. A systematic review of 48 studies including 6,107 cases reported a 17.3% morbidity rate and a 3.7% re-operation rate. Of all complications, postoperative ileus (POI) is the most commonly observed morbidity following ileostomy closure, with rates typically reported between 15-32 %. POI can lead to increased patient discomfort, postoperative morbidity, prolonged hospital stay, increased risk for nosocomial infections,and ultimately higher health care costs.

Transient gut dysmotility can be expected after abdominal surgery. However, in the case of an ileostomy, the defunctionalized segment of bowel undergoes a series of structural and functional changes that may increase the time it takes for motility to resume after closure. Studies performed in animals have shown that defunctionalization of the ileum leads to atrophy of its villi and muscular layers.This was confirmed in humans by Williams et al.,who demonstrated a significant loss of muscular contractility and atrophy of intestinal villi following the creation of a diverting ileostomy.Oh et al. also revealed lower concentrations of peptide YY secreted in the mucosa of the ileum and colon distal to a loop ileostomy,the function of which is to inhibit gastric motility and promote water and electrolyte absorption in the colon.Thus, the absorptive capacity of the colon is reduced following reconstruction of the bowel.

It would appear that changes in the defunctionalized segment of bowel might leave it functionally unprepared for intestinal transit, contributing to the development of POI. A group in Spain proposed that preoperative stimulation of the excluded intestine might reverse those changes and improve its absorptive and motor function prior to restoring intestinal continuity, thus reducing the incidence of POI.They published a randomized controlled trial of 70 patients, of which 35 patients underwent daily stimulation with a thickened saline-based solution via the efferent limb of the ileostomy for two weeks. Following ileostomy closure, they observed reduced rates of POI, earlier return to oral intake and passage of flatus or stool, and shorter hospital stays in the group of patients that underwent stimulation. While their results are promising, t was a single-institution study in a European patient population, perhaps limiting its generalizability to our practice. Furthermore, while randomization should allow for equal distribution of confounders amongst the two groups, they did not report on electrolyte imbalances, narcotic use, and other variables known to influence the development of POI. Miedema and colleagues were the only other group to apply a similar technique of bowel stimulation before ileostomy closure, and found no benefits in intestinal absorptive function or postoperative bowel function. However, they only had six patients in their stimulated group, and all had undergone a restorative proctocolectomy with ileoanal J pouch, thus only a short segment of distal ileum was stimulated.

The idea of stimulating defunctionalized bowel to reduce POI is theoretically plausible, but is lacking in evidence. To our knowledge, this study would be the first of its kind in North America, and would complement the work done in Europe.The potential benefits of this intervention are numerous, including the patient's overall postoperative outcome, a postoperative course with a potential two-day reduction in length of stay and its associated health care costs. If such findings are observed, the use of preoperative bowel stimulation could be incorporated in Enhanced Recovery After Surgery (ERAS®) pathways for patients undergoing ileostomy closure.

The aim of this study is to evaluate the impact of preoperative stimulation of the defunctionalized intestine of a loop ileostomy on postoperative outcomes following ileostomy closure. Investigators hypothesize that preoperative stimulation of the defunctionalized intestine via the efferent limb will reduce the rates of postoperative ileus following ileostomy closure.

This is a multicenter randomized controlled trial involving patients from 4 university hospitals. Patients will be recruited by their individual surgeon, who will explain the objectives of this study and obtain informed consent when obtaining consent for ileostomy closure.

All patients who have undergone an anterior or low-anterior resection for neoplastic (benign and malignant) or diverticular disease with a protective loop ileostomy by a fully trained colorectal/general surgeon or surgical oncologist at one of the involved sites will be offered to enter the study.

Patients with underlying Crohn's disease, with known metastases at the time of ileostomy closure and patients from whom clear and informed consent cannot be obtained will be excluded.

The current overall rate of POI following ileostomy closure at the involved institutions is 16%. Based on the previously published study and the clinical experience, investigators estimate an absolute risk reduction in POI of 13%. With an alpha of 0.05, a power of 0.80 and an estimated 5% loss to follow-up, 83 patients are required in each arm for a total of 166 patients. At each participating institution, at least 35 ileostomy closures eligible for this study are performed per year. Assuming a 70% participation rate, investigators anticipate being able to recruit 122 patients per year for all 5 institutions involved, thus requiring 1.4 years to complete the study. In order to mitigate losses to follow-up, patients will receive a phone call, instructions and equipment for home stimulation if they are unable to come to a stimulation session.

Block randomization will be performed using a computer-generator sequence, to ensure that the initial surgical approach for colorectal resection (open vs. laparoscopic) is equally distributed in the two groups. Group allocation will be concealed from the treating surgeons and researchers involved in the study (except the research assistant doing the stimulation sessions).

All patients enrolled in the study will follow the same preoperative protocol. Upon agreeing to participate in the study, patients will be randomized to either the stimulation group or the non-stimulation (control) group.The protocol for stimulation will be identical for all patients. Stimulation will be performed daily on an outpatient basis for the two weeks (ten business days) prior to ileostomy closure.The efferent limb of the ileostomy loop will be canalized with an 18 Fr Foley catheter and infused with a solution comprising of 500mL of normal saline mixed with 30g of a thickening-agent (Nestle Resource). It will be prepared in five 100mL syringes and administered slowly over 20 minutes.

All surgeries will be performed by an attending colorectal surgeon with the assistance of one or more General Surgery residents. Perioperative antibiotics will include one dose each of cefazolin 1g intravenously and metronidazole 500mg intravenously just prior to surgery. Procedures will be performed under general anesthesia, and a similar operative technique will be used for each case. A parastomal incision will be made and carried out sharply into the peritoneal cavity. Adhesiolysis will be conducted and intestinal continuity will be restored with a side-to-side functional end-to-end enteroenteral stapled anastomosis.The intestine will then be returned to the abdominal cavity. Fascia will be closed with interrupted or running sutures.The fascia will then be infiltrated with 20mL of 0.25% bupivacaine,and the skin will be closed with a purse-string suture and covered by dry dressings.Patients will be given patient-controlled analgesia in the post-anaesthesia care unit for postoperative analgesia. Epidurals will not be used.

Any operation necessitating conversion to a laparotomy incision due to technical difficulties or intraoperative complications will be excluded from analysis.

All patients will follow the perioperative Enhanced Recovery After Surgery (ERAS®) protocol for elective colorectal surgery already implemented at the involved sites. Specifically, this protocol allows for a clear fluid diet on postoperative day 0, and a low-residue diet on the morning of postoperative day 1. If this is well tolerated, the patient is further progressed to a regular diet later in the day. Patients are also encouraged to chew gum and ambulate.

Criteria for granting discharge home from hospital will include the following:

1. tolerating oral diet;
2. no overt abdominal distension;
3. adequate pain control;
4. absence of fever or signs of surgical site infection;
5. ambulating at baseline; and
6. passage of flatus or stool.

Blood work, including CBC and electrolytes (and extended electrolytes), will be drawn daily on postoperative days 1,2, and 3, and then as clinically indicated. All electrolyte abnormalities will be corrected. Nurses will record all narcotic use in patient charts, and this will be converted to morphine equivalents using an equianalgesic table at the time of data collection. A trained, blinded assessor (a physician researcher or colorectal research fellow) will prospectively collect postoperative clinical data by history, physical examination, and chart review. This assessor will be blinded to the stimulation vs. control group assignment and to any preoperative information.

Data regarding patient demographics and specifics of the primary surgery will be collected prospectively, including the indication and approach used for colorectal resection, the length of time between ileostomy creation and closure, and the use of any neoadjuvant or adjuvant treatments in the case of colorectal cancer. All postoperative data will be collected prospectively by the research assistant.

The primary outcome will be postoperative ileus, defined as an intolerance to oral food in the absence of clinical or radiological signs of obstruction, that either a)lasts more than 72 hours; b)requires nasogastric tube insertion; or c)is associated with 2 of the following: nausea/vomiting, abdominal distension, and the absence of flatus. Secondary outcomes will include length of stay, time to tolerating a regular diet, time to first passage of flatus or stool, and overall morbidity. Lastly, an analysis of additional risk factors for postoperative ileus will be performed.

All statistical analyses will be performed using JMP® 11 statistical discovery software (SAS Institute Inc.,Cary,NC,1989-2007). Patient characteristics, clinical variables, POI and other postoperative outcomes will be compared between the two groups using Chi-square, student's t and Wilcoxon rank sum tests for categorical, normally distributed continuous and non-normally distributed continuous variables, respectively. Statistical significance will be considered when p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* All patients will have undergone an anterior or low-anterior resection for malignant or benign disease with a protective loop ileostomy by a board-certified colorectal surgeon or surgical oncologist at one of the involved sites.

Exclusion Criteria:

* Patients with a protective ileostomy following colonic resection for Crohn's disease will be excluded from entering the study, as well as patients from whom clear and informed consent cannot be obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Number of patients with postoperative ileus | Patients will be followed for the duration of hospital stay until discharge, about 30 days
  Number of participants with post-operative ileus lasting longer than 72 hours after loop ileostomy closure and followed up until discharge
Postoperative length of stay | Patients will be followed for the duration of hospital stay until discharge, about 30 days
  (Revised primary outcome: Aug 9th, 2019) Due to slow recruitment, the primary outcome has been changed from postoperative ileus (POI) to postoperative length of stay (LOS). At our institution, the median LOS after loop ileostomy closure among patients managed within an Enhanced Recovery Program was 4.5 days (Garfinkle et al. Br J Surg. 2019). With a standard deviation of 4, the revised power calculations require 63 patients in each arm to identify a reduction in LOS of 2 days with the intervention (Abrisqueta et al. Dis Colon Rectum. 2014) with 80% power and an alpha=0.05. POI will remain a secondary outcome. With the new power analysis, the research team will stop and analyze the data after 126 patients have completed the study follow-up. If at this time there is no difference in LOS between the intervention and control group, the study will continue until the original sample size of 166 patients. This will ensure that the study is powered to detect a difference in both LOS and POI.

CONTACTS AND LOCATIONS:
Overall Officials: Marylise Boutros, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada